CLINICAL TRIAL: NCT05327868
Title: Dietary Inflammation in Older Adults: the Role of Obesity
Brief Title: Lean and Obese: Dietary Inflammation
Acronym: LODI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sue A. Shapses, Ph.D., RD, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2019002228
Record Dates: First submitted 2022-02-28; First posted 2022-04-14 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Inflammation; Dietary Fat
Keywords: obesity; lean individuals; older adults; microbiome; dietary fat
MeSH Terms: conditions — Obesity; Inflammation | interventions — Diet, Fat-Restricted; Diet, High-Fat; Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese (Experimental): BMI in Obesity range
  Interventions: Other: Low Fat Diet (LFD); Other: High Fat Diet (HFD)
- Normal weight (lean) (Experimental): Normal body weight
  Interventions: Other: Low Fat Diet (LFD); Other: High Fat Diet (HFD)

INTERVENTIONS:
Other: Low Fat Diet (LFD) — Subjects will be asked to adhere to a low fat diet (assigned in random order) and be counseled by a dietitian using 5 days of sample menus, monitored online using a shared nutrient analysis program, and supplied with low fat foods to increase compliance
  Other Names: low fat diet
Other: High Fat Diet (HFD) — Subjects will be asked to adhere to a high fat diet that is rich in SFAs (assigned in random order) and be counseled by a dietitian using sample 5 days of menus, monitored online using a shared nutrient analysis program, and supplied with high fat foods to increase compliance
  Other Names: high fat (high SFA) diet

SUMMARY:
In the Lean and Obese Dietary Inflammation (LODI) study, the primary goal is to determine the effect of short-term intake of high dietary fat (5 days) compared to low fat intake (5 days) in a cross-over design in older adults (men and women) with normal body weight or obesity. Inflammation will be examined by measuring serum endotoxin and other markers, as well as the fecal microbiota.

DETAILED DESCRIPTION:
In the Lean and Obese Dietary Inflammation (LODI) study, short-term intake of a high-fat diet (HFD) that is also high in saturated fatty acids will be examined compared to a low-fat diet (LFD) in individuals who are normal body weight (BMI 19.5-24.9) or who have obesity (BMI of 30 - 40 kg/m2). To characterize persons at baseline, this study will examine body composition, and serum glucose, endotoxin, inflammation and intestinal permeability during fasting and in response to a mixed meal. Also, while it is known that long term intake of foods affects the microbiota, it is unclear whether short-term consumption of a HFD will shift towards a pro-inflammatory gut microbiota compared to a low fat intake. This will be tested in a cross-over design (5 days on a HFD, washout, and 5 days on a LFD) with order randomly assigned in older adults (50+ years of age) who have obesity or are normal weight, and will also be examined by estimated visceral adipose tissue level.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women
* Age 50-79 years (only postmenopausal women > 2 years)
* Body mass index (20-25 kg/m2; and 30-40 kg/m2)*

Exclusion Criteria:

* Diagnosed with, active, or history of liver cirrhosis, chronic or persisting hepatitis
* Diagnosed with, active, or history of cancer
* History of gastrointestinal disease or surgical procedure for weight loss.
* Diagnosed with immune diseases, type 2 diabetes, pancreatitis, or infectious diseases
* Any surgery in the past 6 months
* Currently using or have used antibiotics continuously > 3 days in the past 3 months
* Regular use of medications for that affect the gastrointestinal tract, cholecystitis, urinary tract infection, severe organic diseases including coronary heart disease, myocardial infarction, infectious diseases including pulmonary tuberculosis and AIDS
* Known allergy or intolerance to any ingredients in the dietary intervention program
* Alcohol or illicit drug abuse
* Current Smoker or have quit smoking in the past 3 months
* Recent colonoscopy (within the previous two months)
* Inability to follow any of the experimental diets (including low or high fat diet) or to perform the collections required for this study
* Participants will also be excluded if they have extreme dietary habits, extreme levels of physical or athletic activity, or by changes in body weight >5 lbs. during the last 6 months
* Uncontrolled hypertension or uncontrolled hyperlipidemia in abnormal ranges.
* Participation in another clinical research trial that may interfere with the results of this study.

  * As needed, BMI (kg/m2) will be adjusted accordingly for Asian lean and obese definitions

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
Change in Endotoxin from Low to High fat diet | Change from LFD (5 days) to HFD (5 days) over an average of 6 weeks
  serum and stool
Change in Microbiome composition | Change from LFD (5 days) to HFD (5 days) over an average of 6 weeks
  stool

SECONDARY OUTCOMES:
Inflammatory markers | Change from LFD (5 days) to HFD (5 days) over an average of 6 weeks
  Serum IL-6, hsCRP, TNF-alpha, TLR4 (grams/volume)
Zonulin | Change from LFD (5 days) to HFD (5 days) over an average of 6 weeks
  Serum
Lipopolysaccharide binding protein (LBP) | Change from LFD (5 days) to HFD (5 days) over an average of 6 weeks
  Serum
Toll like receptor-4 and Null 2 stimulation | Change from LFD (5 days) to HFD (5 days) over an average of 6 weeks
  serum and the HEK cell reporter assay
Endotoxin in response to a meal | Change over 5 hour MMT
  Serum inflammatory response to a mixed meal tolerance test (MMT)

OTHER OUTCOMES:
Change in Glucose in response to a meal | Change over 5 hour MMT
  Serum glycemic response to a meal
Change in insulin in response to a meal | Change over 5 hour MMT
  Serum glycemic response to a meal
Inflammatory markers in response to a meal | Change over 5 hour MMT
  serum TNF alpha, CRP and IL-6 (grams/volume)
Lipopolysaccharide binding protein (LBP) in response to a meal | Change over 5 hour MMT
  serum
Change in Triglycerides in response to a meal | Change over 5 hour MMT
  Serum lipid response to a meal (peak and AUC)
Change in Osteocalcin in response to a meal | Change over 5 hour MMT
  Serum bone formation and energy metabolism marker
Change in PINP in response to a meal | Change over 5 hour MMT
  Serum bone formation marker
Change in CTX in response to a meal | Change over 5 hour MMT
  Serum bone resorption marker
Change in diet quality score | Change from LFD (5 days) to HFD (5 days) over an average of 6 weeks
  Nutrient analysis and HEI (higher score is better)
Body composition in lean and obese weight groups | baseline characteristics
  total tissue, fat-free soft tissue, fat, visceral adiposity

CONTACTS AND LOCATIONS:
Overall Officials: Sue Shapses, PhD, Principal Investigator — Rutgers, the State University
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results and after deidentification will be shared upon request for researchers who provide a methodologically sound proposal (and IRB approved).

REFERENCES:
- [Derived] Ogilvie AR, Onishi JC, Schlussel Y, Kumar A, Haggblom MM, Kerkhof LJ, Shapses SA. Short-term high fat diet-induced metabolic endotoxemia in older individuals with obesity: a randomized crossover study. Am J Clin Nutr. 2025 Aug;122(2):601-611. doi: 10.1016/j.ajcnut.2025.06.001. Epub 2025 Jun 4. PMID 40480607

DOCUMENTS (1):
  • Informed Consent Form (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT05327868/ICF_000.pdf